CLINICAL TRIAL: NCT03069274
Title: Impact of a Randomized School-based Intervention on Sugar-sweetened Beverage Intake Substitution by Water to Prevent Excessive Weight in Mexican Scholars
Brief Title: Sugar-sweetened Beverage Intake Substitution by Water to Prevent Overweight in Mexican Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, LILIA CASTILLO MARTINEz, Medical Rearch Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NC001
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Only general nutritional recommendations were given.
  Interventions: Behavioral: General nutritional recommendations
- Intervention (Experimental): General nutritional recommendations, change their drinking habits.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — General nutritional recommendations, change drinking habits
  Other Names: General nutritional recommendations, change drinking habits
  Arms: Intervention
Behavioral: General nutritional recommendations — Only general nutritional recommendations were given
  Arms: Control

SUMMARY:
The prevalence of overweight and obesity in children have increased in recent years and this has been associated with replacing plain water intake by sugar-sweetened beverages.

Because of this, the objective of the present study was to evaluate the impact of a school-based intervention that aimed to replace sugar-sweetened beverages by water.

A randomized community trial including 314 children aged 9-11 years from three public schools of the State of Hidalgo, Mexico was performed. Schools were randomized to intervention (two schools from municipality of Apan; six classes with 146 participants) or control group (one school from municipality of Emiliano Zapata; six classes with 168 participants) and followed during 6 months. Intervention included to place water filters at school and classroom lessons to increase water consumption and decreasing sugar-sweetened beverages.

DETAILED DESCRIPTION:
This was a randomized community trial, that included children of both sexes belonging to public elementary schools, grades 4 and 5, in Hidalgo, Mexico, including the municipalities of Emiliano Zapata and Apan. It was excluded from school children with Type 1 Diabetes, heart failure, kidney or liver that limit fluid intake by medical prescription.

A sample size of 334 (167 in each group) children would allow to detect a difference of 9% in water consumption between the two groups15, considering a loss to follow-up of 20%, a power of 85% and a significance level of 0.05.

The selection of the schools of the two communes was based on the availability of a place to conduct physical assessments and intervention. Schools were randomly assigned to the intervention (IG) or control groups (CG). Each group included 3 classes of fourth grade and 3 classes of fifth grade.

Written informed consent was obtained from school principals, teachers, parents and students. The study was approved by the Ethics Committee of the Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubiran, in Mexico City.

Measurements Study variables were measured at baseline and at 6 months after intervention. Weight was measured with a portable scale (SECA professional scale model 750, Seca North America East, Hanover, MD) with a capacity of 150 kg and a precision of 1kg, height (SECA model 280 portable stadiometer, Seca North America East, Hanover, MD) with an amplitude of 220 cm and variation of 1 mm. Subjects were weighed and measured with minimal clothing and no shoes21. Body mass index (BMI) was calculated as weight (in kg) divided by stature2 (in m). Classification of nutritional status was based on z-scores of the BMI-for-age and sex from the distributions of the World Health Organization using the Anthro-Plus software22.

Body composition was evaluated by bioelectric impedance, using multiple frequency equipment (RJL Systems, Detroit, MI). Resistance and reactance were obtained to estimate body fat and fat-free mass were estimated using equations23.

Sugar-sweetened beverage and water plain consumption were measured at the beginning and end of the study through a 24-hour recall using ESHA Food software with an SQL processor (version 7.9, ESHA Research, Salem, OR, 2001)., with face-to-face interviews in each phase.

Intervention The intervention focused on encouraging students to change their drinking habits over 6 months (from January to June) in the school year of 2015.

In the intervention group, reusable plastic water bottles and jugs were delivered at school and water filters were placed. Classroom lessons lasting 30 minutes were conducted weekly by trained nutritionists. These sessions included general nutritional recommendations, encouragement of simple water plain consumption and discouragement of consumption of sugar-sweetened beverages, through a manual of drinks, developed by nutritionists. In the control group only general nutritional recommendations were given.

ELIGIBILITY:
Inclusion Criteria:

* Children 8-12 years old
* Both sexes
* Belonging to public elementary schools, grades 4 and 5, in Hidalgo, Mexico

Exclusion Criteria:

* Type 1 Diabetes
* Heart kidney or liver failure
* Limitation of fluid intake by medical prescription.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 314 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-11-08 (Actual)

PRIMARY OUTCOMES:
Change their drinking habits | Baseline and 6 months follow up
  Decrease sugar-sweetened beverage and increase water plain consumption evaluating the change at the beginning and end of the study through a 24-hour recall using ESHA Food software with an SQL processor with face-to-face interviews in each phase.

CONTACTS AND LOCATIONS:
Overall Officials: LILIANA RUIZ-ARREGUI, PhD, Study Chair — INSTITUTO NACIONAL DE CIENCIAS MEDICAS Y NUTRICION SZ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barquera S, Campirano F, Bonvecchio A, Hernandez-Barrera L, Rivera JA, Popkin BM. Caloric beverage consumption patterns in Mexican children. Nutr J. 2010 Oct 21;9:47. doi: 10.1186/1475-2891-9-47. PMID 20964842
- [Background] Malik VS, Popkin BM, Bray GA, Despres JP, Willett WC, Hu FB. Sugar-sweetened beverages and risk of metabolic syndrome and type 2 diabetes: a meta-analysis. Diabetes Care. 2010 Nov;33(11):2477-83. doi: 10.2337/dc10-1079. Epub 2010 Aug 6. PMID 20693348
- [Background] Nissinen K, Mikkila V, Mannisto S, Lahti-Koski M, Rasanen L, Viikari J, Raitakari OT. Sweets and sugar-sweetened soft drink intake in childhood in relation to adult BMI and overweight. The Cardiovascular Risk in Young Finns Study. Public Health Nutr. 2009 Nov;12(11):2018-26. doi: 10.1017/S1368980009005849. Epub 2009 May 28. PMID 19476678
- [Background] Hoelscher DM, Kirk S, Ritchie L, Cunningham-Sabo L; Academy Positions Committee. Position of the Academy of Nutrition and Dietetics: interventions for the prevention and treatment of pediatric overweight and obesity. J Acad Nutr Diet. 2013 Oct;113(10):1375-94. doi: 10.1016/j.jand.2013.08.004. PMID 24054714
- [Background] Kenney EL, Gortmaker SL, Carter JE, Howe MC, Reiner JF, Cradock AL. Grab a Cup, Fill It Up! An Intervention to Promote the Convenience of Drinking Water and Increase Student Water Consumption During School Lunch. Am J Public Health. 2015 Sep;105(9):1777-83. doi: 10.2105/AJPH.2015.302645. Epub 2015 Jul 16. PMID 26180950